CLINICAL TRIAL: NCT03643692
Title: Adaptive, Real-time, Intelligent System to Enhance Self-care of Chronic Disease
Acronym: ARISES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18HH4410
Record Dates: First submitted 2018-08-13; First posted 2018-08-23 (Actual); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus; blood glucose; environmental case parameters
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARISES (Experimental): Observational study using wearable technologies to collect data and evaluate blood glucose correlations against physiological and environmental case parameters. Useful associations will assist the development of the CBR/machine learning algorithm and identify wearable devices for the final ARISES platform.
  Interventions: Device: ARISES

INTERVENTIONS:
Device: ARISES — The Adaptive, Real-time, Intelligent System to Enhance Self-care of chronic diseases (ARISES) project will use type 1 diabetes (T1DM) as an exemplary case study to demonstrate safety, technical proof of concept and efficacy of a novel mobile platform. Combining wearable sensors and smartphone technology, a range of biological, environmental and behavioural data will be analysed to provide real-time therapeutic and lifestyle decision support. Using Case-Based-Reasoning (CBR), the system will be adaptive and personalised with the ability to learn from previously encountered scenarios. Ultimately, ARISES aims to empower self-management of chronic illness and limit the complications associated suboptimal treatment.

SUMMARY:
The Adaptive, Real-time, Intelligent System to Enhance Self-care of chronic diseases (ARISES) project will use type 1 diabetes (T1DM) as an exemplary case study to demonstrate safety, technical proof of concept and efficacy of a novel mobile platform. Combining wearable sensors and smartphone technology, a range of biological, environmental and behavioural data will be analysed to provide real-time therapeutic and lifestyle decision support. Using Case-Based-Reasoning (CBR), the system will be adaptive and personalised with the ability to learn from previously encountered scenarios. Ultimately, ARISES aims to empower self-management of chronic illness and limit the complications associated suboptimal treatment.

DETAILED DESCRIPTION:
ARISES will target self-management to optimise glucose control through insulin dose recommendation (therapeutic advice), exercise and stress support, hypoglycaemia prevention through timely snack recommendation and behavioural change through educational support (lifestyle advice).

Semi-structured focus meetings comprised of patients with T1DM, clinicians, engineers and experts in human-computer interaction will provide a forum to establish the essential usability requirements to incorporate into the ARISES mobile interface. The design will focus on ensuring access to decision support is intuitive and efficient while maintaining sight of real-time glycaemia outcomes. The design and implementation of the user-interface will be assessed in a series of usability validation studies.

Clinical studies will be conducted in two phases. The first phase will be an observational study using wearable technologies to collect data and evaluate blood glucose correlations against physiological and environmental case parameters. Useful associations will assist the development of the CBR/machine learning algorithm and identify wearable devices for the final ARISES platform.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18years of age
* Diagnosis of T1DM for > 1 year
* Structured education completed in last 3 years and capable of CHO counting
* CBG measured at least twice daily for CGM calibration
* Capacity to follow the protocol and sign the informed consent
* Access to a personal computer/laptop

Exclusion Criteria:

* Severe episode of hypoglycaemia (requiring 3rd party assistance) in last 6 months
* Diabetic ketoacidosis in the last 6 months prior to enrolment
* Impaired awareness of hypoglycaemia (based on Gold score)
* Pregnant or planning pregnancy over time of study procedures
* Breastfeeding
* Enrolled in other clinical trials
* Active malignancy or being investigated for malignancy
* Suspected or diagnosed endocrinopathy like adrenal insufficiency, unstable thyroidopathy, endocrine tumour
* Gastroparesis
* Autonomic neuropathy
* Macrovascular complications (acute coronary syndrome, transient ischaemic attack, cerebrovascular event within the last 12 months prior to enrolment in the study)
* Visual impairment including unstable proliferative retinopathy
* Reduced manual dexterity
* Inpatient psychiatric treatment
* Abnormal renal function test results (calculated GFR <40 mL/min/1.73m2)
* Liver cirrhosis
* Not tributary to optimization to insulin therapy
* Abuse of alcohol or recreational drugs
* Oral steroids
* Regular use of the paracetamol, beta-blockers or any other medication that the investigator believes is a contraindication to the participant's participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ARISES: ARISES: The Adaptive, Real-time, Intelligent System to Enhance Self-care of chronic diseases (ARISES) project will use type 1 diabetes (T1DM) as an exemplary case study to demonstrate safety, technical proof of concept and efficacy of a novel mobile platform. Combining wearable sensors and smartphone technology, a range of biological, environmental and behavioural data will be analysed to provide real-time therapeutic and lifestyle decision support. Using Case-Based-Reasoning (CBR), the system will be adaptive and personalised with the ability to learn from previously encountered scenarios. Ultimately, ARISES aims to empower self-management of chronic illness and limit the complic
Period: Overall Study
Arm/Group | ARISES
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ARISES
Number analyzed (Participants) | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [28 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Insulin Modality: Insulin pump (CSII), Multiple daily injections (MDI) [Count of Participants; unit: Participants]
  CSII | 6
  MDI | 6

OUTCOME MEASURES:

1. Primary Outcome: Time in Range (%)
Description: % time in target range (3.9 - 10 mmol/L) without insulin dose increase
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time (minutes)
Arm/Group | ARISES
Number analyzed (Participants) | 12
percentage of time (minutes) | 64 [54.4 to 77.3]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | ARISES
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARISES (N=12)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Rash from empatica watch

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT03643692/Prot_SAP_000.pdf